CLINICAL TRIAL: NCT06364241
Title: Focus Groups on Cognitive Function in Psychosis
Acronym: PRECOGNITION
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 331760; 226706/Z/22/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2024-03-18; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Psychosis
Keywords: Schizophrenia; Bipolar disorder; Cognition
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Bipolar Disorder | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with lived experience of psychosis: Individuals with lived experience of psychosis
  Interventions: Other: Focus group
- Carers of individuals with lived experience of psychosis: Carers of individuals with lived experience of psychosis
  Interventions: Other: Focus group

INTERVENTIONS:
Other: Focus group — During the focus group, the investigators will explore the cognitive deficits that people with lived experience with psychosis and their carers consider to be the most impairing.

SUMMARY:
Cognitive deficits are commonly observed in people with mental disorders. In psychosis, these impairments are frequently present early in the course of the disorder and have a substantial impact on functional outcomes. This project will gain insight into the cognitive deficits that people with lived experience of psychosis and their carers perceive to be the most troublesome. To achieve this, the investigators will conduct two sets of focus groups. During the first set of focus groups, the investigators will aim to identify the cognitive deficits that individuals with psychosis and their carers consider to be the most impairing.

The findings of these focus groups will provide important information about what areas of cognition and functioning should be considered in future analyses of large fully anonymised datasets collected in the past from individuals with psychosis. The focus groups will not form part of those analyses, but will provide input from people with lived experience of psychosis on what problems with thinking skills are the most important for them and that should be considered by further research.

The second set of focus groups will enable the investigators to determine the participants' perception of potential risks and benefits associated with the dissemination of findings on cognitive function in psychosis, to ensure this is done in a manner that is sensitive to the wishes and needs of people with lived experience of psychosis.

Each participant will be asked to attend one focus group, which will last approximately one hour. Focus groups will take place at the South London and Maudsley (SLaM) Trust or at the Institute of Psychiatry, Psychology and Neuroscience (IoPPN), King's College London, although provision will be made for participants to also participate online.

DETAILED DESCRIPTION:
Design The investigators will conduct two sets of focus groups (2 focus groups at the beginning and 1 or 2 focus groups at the end of the project) with a total of 6-8 participants each. Focus groups will include either with people with lived experience with psychosis or carers of people with lived experience with psychosis.

Timetable Attempts to contact participants will begin as soon as ethical approvals are in place. It is expected that data collection will be completed over a 4-6-month period. Interpretation and analysis of findings and preparation of the final report will be completed by 30/09/2026.

Methodology Each focus group will last approximately one hour and will be conducted by a research group member with relevant expertise. The focus groups will be held in-person at the Institute of Psychiatry, Psychology and Neuroscience (IoPPN) Main Building, King's College London, although provision will be made for participants to also participate online via Microsoft Teams. The focus groups will be conducted in close temporal proximity one to another. The focus groups will be facilitated by project staff, including project members with lived experience of psychosis. Participants will be reimbursed for their time in participating in the focus groups and for their travel expenses to attend. The focus groups will be recorded (audio only) with participants' informed consent. Focus group data will be transcribed verbatim by a professional transcription company.

The first set of focus groups will explore the cognitive deficits that people with lived experience of psychosis or their carers consider to be the most impairing. The second set of focus groups will discuss the results that emerge from this project, paying particular attention to the participants' views on both the risks and potential opportunities derived from our project, including recommendations regarding future stages of research. The investigators will also discuss the best way to present findings to the wider scientific community and lay audiences.

For each set of focus groups, thematic analysis will be conducted to order data into meaningful patterns. Thematic analysis will include inductive and deductive coding to ensure that analysis is shaped by participants' concerns and priorities, and allow the investigators to systematically probe the data, asking questions arising from the existing literature. Thematic analysis will be performed using the Atlas.ti software, which is an industry standard for both deductive and inductive analyses. Finally, the findings from the focus groups will be disseminated via publications prepared with input from the lived experience experts.

ELIGIBILITY:
Inclusion Criteria:

* Lived experience with psychosis, including individuals with personal experience of psychosis, carers and family members
* Current or past cognitive deficits
* Age between 18 and 65 years
* Able to provide informed consent

Exclusion Criteria:

* No lived experience with psychosis
* Traumatic brain injury
* Neurological or metabolic disorders associated with cognitive deficits
* On occasions where it is not possible for the protocol to be followed, i.e. due to language barriers, participants will not be consented into the study

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals with lived experience with psychosis, including individuals with personal experience of psychosis, carers and family members
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Individual perception of impairments due to cognitive deficits associated with psychosis | Autumn 2024
  For each set of focus groups, thematic analysis will be conducted to identify the main cognitive deficits that people with lived experience with psychosis consider to be the most impairing, including deficits in working memory, executive function and attention. No structured scales or questionnaires will be used.

IPD SHARING:
Plan to Share IPD: No